CLINICAL TRIAL: NCT05746559
Title: ARTEMIS: RAvulizumab to PRotect PaTients With Chronic Kidney DisEase (CKD) froM Cardiac Surgery Associated Acute Kidney Injury (CSA-AKI) and Subsequent Major Adverse Kidney Events (MAKE): A Phase 3, Randomized, Double-blind, Placebo-controlled, Multicenter Study
Brief Title: ARTEMIS: Ravulizumab to Protect Patients With CKD From CSA-AKI and MAKE
Acronym: ARTEMIS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D928DC00001; ALXN1210-CSA-AKI-318 (Other: Alexion Pharmaceuticals, Inc.); 2022-501802-36 (EudraCT Number)
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Chronic Kidney Disease; CKD; Cardiac Disease; Cardiopulmonary Bypass
Keywords: Chronic Kidney Disease; CKD; Cardiac Disease; Cardiopulmonary Bypass
MeSH Terms: conditions — Renal Insufficiency, Chronic; Heart Diseases | interventions — ravulizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive a single weight-based dose of placebo via intravenous infusion, 1 to 7 days prior to surgery.
  Interventions: Drug: Placebo
- Ravulizumab (Experimental): Participants will receive a single weight-based dose of ravulizumab, via intravenous infusion, 1 to 7 days prior to surgery.
  Interventions: Drug: Ravulizumab

INTERVENTIONS:
Drug: Placebo — Participants will receive a single weight-based dose of placebo via intravenous infusion.
  Arms: Placebo
Drug: Ravulizumab — Participants will receive a single weight-based dose of ravulizumab via intravenous infusion.
  Arms: Ravulizumab

SUMMARY:
The primary objective of this study is to assess the efficacy of a single dose of ravulizumab IV compared with placebo in reducing the risk of the clinical consequences of AKI (MAKE) at 90 days in adult participants with CKD who undergo non-emergent cardiac surgery with CPB.

ELIGIBILITY:
Inclusion Criteria:

* Participant weighs ≥ 30 kg
* Planned non-emergent sternotomy with CPB procedure for the following surgeries:
* Multi-vessel CABG
* Valve replacement or repair; ascending aorta surgery permitted if combined with aortic valve replacement/repair
* Combined CABG and valve surgery; inclusion of single-vessel CABG when combined with valve replacement/repair is permitted
* Known CKD for at least 90 days (CKD Stage 3A, 3B, or 4)

Exclusion Criteria:

* Emergency or salvage cardiac surgery is expected at screening or randomization, as assessed by the investigator.
* Single-vessel CABG without valve surgery is planned.
* Off-pump surgery is planned (eg, surgery without CPB).
* Recipient of a solid organ or bone marrow transplantation.
* Cardiogenic shock, hemodynamic instability, use of intra-aortic balloon pump, extracorporeal membrane oxygenation, or left ventricular assist device within 72 hours of randomization.
* Active systemic bacterial, viral, or fungal infection within 14 days prior to randomization.
* History of unexplained, recurrent infection.
* Any use of KRT or presence of AKI within 30 days of randomization
* Use of any complement inhibitors, or plasmapheresis or plasma exchange within the year prior to Screening, or planned use during the course of the study.
* Participant is not willing to be vaccinated against N meningitidis or is unwilling to receive prophylactic treatment with appropriate antibiotics , if needed
* History of or unresolved N meningitidis infection.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 736 (Estimated)
Dates: Start 2023-04-06 (Actual); Primary Completion 2026-05-18 (Estimated); Study Completion 2027-02-17 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Major Adverse Kidney Events (MAKE) (Based on serum Cystatin C [sCysC]) at Day 90 Post Cardiopulmonary Bypass (CPB) | Day 90 post-CPB

SECONDARY OUTCOMES:
To assess the efficacy of ravulizumab in reducing risk of AKI (based on sCr) following CPB | Day 90 post CPB
  1. Occurrence of CSA-AKI without recovery at Day 90 post CPB
  2. Occurrence of severe CSA-AKI (KDIGO Stage 2 or 3) from randomization to Day 7 post CPB
  3. Occurrence of severe AKI (KDIGO Stage 2 or 3) from randomization to Day 30 post CPB
  4. Occurrence of KRT or death from randomization to Day 90 post CPB
  5. All-cause mortality from randomization to Day 90 post CPB
  6. Length of post-operative ICU stay

CONTACTS AND LOCATIONS:
Locations (139):
- United States (28):
  - Research Site, Tucson, Arizona
  - Research Site, Orange, California
  - Research Site, San Francisco, California
  - Research Site, Stanford, California
  - Research Site, Aurora, Colorado
  - Research Site, Weston, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Boston, Massachusetts
  - Research Site, Springfield, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Rochester, New York
  - Research Site, Valhalla, New York
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Dallas, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Charlottesville, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Seattle, Washington
- Argentina (4):
  - Research Site, Buenos Aires
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Corrientes
  - Research Site, Santa Fe
- Australia (5):
  - Research Site, Adelaide
  - Research Site, Brisbane
  - Research Site, Monash
  - Research Site, Murdoch
  - Research Site, Southport
- Research Site, Vienna, Austria
- Brazil (9):
  - Research Site, Belo Horizonte
  - Research Site, Brasília
  - Research Site, Fortaleza
  - Research Site, Recife
  - Research Site, Ribeirão Preto
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Canada (7):
  - Research Site, Edmonton, Alberta
  - Research Site, Winnipeg, Manitoba
  - Research Site, Saint John, New Brunswick
  - Research Site, Hamilton, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- China (8):
  - Research Site, Beijing
  - Research Site, Huai'an
  - Research Site, Shanghai
  - Research Site, Shenzhen
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Zhengzhou
- France (4):
  - Research Site, Bordeaux
  - Research Site, Dijon
  - Research Site, Montpellier
  - Research Site, Toulouse
- Germany (9):
  - Research Site, Essen
  - Research Site, Frankfurt am Main
  - Research Site, Giessen
  - Research Site, Halle
  - Research Site, Heidelberg
  - Research Site, Jena
  - Research Site, München
  - Research Site, Stuttgart
  - Research Site, Trier
- Research Site, Hong Kong, Hong Kong
- India (6):
  - Research Site, Bangalore
  - Research Site, Delhi
  - Research Site, Gūrgaon
  - Research Site, Hyderabad
  - Research Site, Mysuru
  - Research Site, Secunderabad
- Research Site, Haifa, Israel
- Italy (4):
  - Research Site, Bari
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Napoli
- Japan (9):
  - Research Site, Bunkyō City
  - Research Site, Chūōku
  - Research Site, Kamakura-shi
  - Research Site, Kawasaki-shi
  - Research Site, Minatoku
  - Research Site, Okayama
  - Research Site, Sagamihara-shi
  - Research Site, Suginami City
  - Research Site, Urayasu
- Netherlands (2):
  - Research Site, Groningen
  - Research Site, Maastricht
- Poland (10):
  - Research Site, Bialystok
  - Research Site, Bielsko-Biala
  - Research Site, Chrzanów
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Poznan
  - Research Site, Szczecin
  - Research Site, Tychy
  - Research Site, Warsaw
- South Korea (6):
  - Research Site, Anyang-si
  - Research Site, Bucheon-si
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (9):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Navarra
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Valladolid
- Taiwan (6):
  - Research Site, Hualien City
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
- Turkey (Türkiye) (5):
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Istanbul
  - Research Site, Menemen/Izmir
  - Research Site, Odunpazari
- United Kingdom (5):
  - Research Site, Cambridge
  - Research Site, Clydebank
  - Research Site, Edinburgh
  - Research Site, London
  - Research Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Derived] Ostermann M, Corteville DC, Doi K, Koyner JL, Lamy A, Li G, Solinsky CM, Winterberg PD, Smith WT, Mehta RL, Murray PT, Shaw AD, Zarbock A, Engelman DT. A phase 3 study of ravulizumab to protect patients with chronic kidney disease from cardiac surgery-associated acute kidney injury and major adverse kidney events (ARTEMIS). Trials. 2025 May 30;26(1):181. doi: 10.1186/s13063-025-08895-7. PMID 40448185